CLINICAL TRIAL: NCT02100618
Title: Evaluation of Antibody Persistence for GSK Biologicals' HPV-16/18 L1 VLP AS04 Vaccine (GSK-580299) Administered in Healthy Adults and Adolescents, 6.5 Years After First Vaccination in the Primary Study
Brief Title: Antibody Persistence for GlaxoSmithKline (GSK) Biologicals' HPV-16/18 L1 VLP AS04 Vaccine (GSK-580299) Administered in Healthy Adults and Adolescents, 6.5 Years After First Vaccination in the Primary Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to late study start, the possibility to enroll enough subjects dropped below the limit to provide scientifically acceptable data, hence study was cancelled.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200255; 2014-000060-17 (EudraCT Number)
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Infections, Papillomavirus
Keywords: Adolescents; Adults; Immunogenicity; 6.5 years; Safety; Antibody persistence; Human Papillomavirus (HPV) vaccine
MeSH Terms: conditions — Papillomavirus Infections | interventions — Blood Specimen Collection; human papillomavirus vaccine, L1 type 16, 18

ARMS (2):
- HPV Group 1 (Experimental): Subjects who were aged 9-14 years at study entry and received two doses of the HPV-16/18 vaccine according to a 0,6-months schedule in the study HPV-048 PRI (NCT00541970).
  Interventions: Procedure: Blood sampling
- HPV Group 2 (Active Comparator): Subjects who were aged 15-25 years at study entry and received three doses of the HPV 16/18 vaccine according to a 0,1,6-months schedule in the study HPV-048 PRI (NCT00541970).
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Blood samples will be collected from all subjects at Year 6.5
  Other Names: Cervarix™

SUMMARY:
The purpose of this study is to establish the long-term persistence of the immune response and safety of the HPV vaccine in healthy females who were aged 9 to 25 years in the primary study (NCT00541970).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol or subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* Subjects who completed their primary vaccination and received either two or three doses of GSK Biologicals' HPV-16/18 vaccine according to a 0,6-months schedule or a 0,1,6-months schedule in the study HPV-048 PRI (110659) (NCT00541970).
* A female between, and including, 9 and 14 years of age or 15 and 25 years of age, at the time of first vaccination, depending on which group they belonged to in the study HPV-048 PRI (110659) (NCT00541970), i.e., 9-14 year old subjects should have received two doses of GSK Biologicals' HPV-16/18 vaccine according to a 0,6-months schedule and 15-25 year old subjects should have received three doses of GSK Biologicals' HPV-16/18 vaccine according to a 0,1,6-months schedule.
* Written informed consent obtained from the subject/from the parent(s)/LAR(s) of the subject. In addition, subjects below the legal age of consent should sign and personally date a written informed assent form.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the HPV-16/18 study vaccine administered in the study HPV-048 PRI (110659) (NCT00541970) from the last visit of the primary study up to the current study visit or planned use during the study period.
* Administration of any HPV vaccine from the last visit of the primary study up to the current study visit or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within three months prior to blood sampling. Inhaled and topical steroids are allowed.
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before study entry, with the exception of routine meningococcal, inactivated influenza, hepatitis B, diphtheria/tetanus and/or diphtheria/tetanus-containing, poliomyelitis and/or pertussis vaccines up to 8 days before study entry. Enrolment will be deferred until the subject is outside of specified window.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Cancer or autoimmune disease under treatment.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the blood sampling.

Ages: 15 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of immune persistence in terms of antibody titres | 6.5 years after first vaccination with HPV-16/18 administered in the study HPV-048 PRI (NCT00541970)

SECONDARY OUTCOMES:
Evaluation of immunogenicity in terms of seroconversion rates (SCRs) and antibody titres | 6.5 years after first vaccination with HPV-16/18 (20 µg of each antigen) administered in the study HPV-048 PRI (NCT00541970)
Occurrence of SAEs | After primary study completion (Month 60) up to end of the study (Visit 1 at Year 6.5)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline